CLINICAL TRIAL: NCT04107961
Title: A Phase II Study to Assess the Safety and Efficacy of the Leishmania Vaccine ChAd63-KH for the Prevention of Post-kala Azar Dermal Leishmaniasis
Brief Title: A Study to Assess Safety and Efficacy of a Leishmania Vaccine to Prevent Post Kala Azar Dermal Leishmaniasis (PKDL)
Acronym: LEISH3
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial will be undertaken but the protocol will be substantially revised.
Sponsor: University of York (Other)
Collaborators: Wellcome Trust (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); European Vaccine Initiative (Other)
Responsible Party: Principal Investigator, Paul Kaye, Project Lead, University of York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LEISH3 (RIA2016V-1640)
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Post-kala-azar Dermal Leishmaniasis
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine arm (Experimental): Vaccine in 1 ml, single dose
  Interventions: Biological: Vaccine
- Placebo (Placebo Comparator): 1 ml normal saline , single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Vaccine — Single intramuscular injection into the deltoid region
  Other Names: ChAd63-KH
  Arms: Vaccine arm
Other: Placebo — Single intramuscular injection into the deltoid region
  Arms: Placebo

SUMMARY:
The actual format of the anticipated LEISH3 trial is under review.

DETAILED DESCRIPTION:
The leishmaniases are poverty-related neglected diseases with a major impact on health worldwide. They affect the poorest of the poor and present a severe barrier to socio-economic development. Caused by infection with one of several species of Leishmania parasite, these diseases occur in 98 countries worldwide and can be broadly classified as tegumentary leishmaniases (TL; affecting the skin and mucosa) and visceral leishmaniasis (VL; affecting internal organs). Worldwide, over 1 million reported cases of TL and 0.5 million reported cases of VL occur each year. Whereas TL are chronic and non-life-threatening, VL is responsible for over 20,000 deaths per year, second only to malaria amongst parasites with regard to mortality. Collectively, approximately 2.4 million disability-adjusted life years are lost to the leishmaniases. No vaccines are currently licensed for any form of human leishmaniasis and the drug arsenal is limited and increasingly compromised by drug resistance.

.

ELIGIBILITY:
Inclusion Criteria:

The patient volunteer must be:

* Aged 12 to 50 years on the day of screening
* Have had VL and have been cured following a standard regimen of SSG / PM
* Females must be unmarried, single, or widowed
* Willing and able to give written informed consent
* For adolescents aged 12 to 17 years on the day of screening written informed consent from a parent must be obtained.

All Participants

* Uncomplicated VL responsive to SSG / PM treatment
* Have relatively normal blood values in the setting of VL, defined as hemoglobin >5.0 g/dL, white blood cells >1.0 x10(9)/L, platelets >40 x10(9)/L, liver function tests < x5 normal, Creatinine <1.5 mg/dL
* Available for the duration of the study
* Without any other significant health problems as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Negative for malaria on blood smear
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol
* Negative for human immunodeficiency virus (HIV), Hepatitis B and Hepatitis C
* For females only, willing to undergo urinary pregnancy tests on the day of screening, on the day of vaccination (prior to vaccination) and 3, 6, 9 and 12 months after vaccination.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Has HIV/VL coinfection
* Has had previous treatment for VL with relapse
* Receipt of a live attenuated vaccine within 60 days or other vaccine within 14 days of screening
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or a history of severe or multiple allergies to drugs or pharmaceutical agents
* Any history of severe local or general reaction to vaccination as defined as
* Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
* General: fever ≥ 39.5°C within 48 hours, anaphylaxis, bronchospasm, laryngeal oedema, collapse, convulsions or encephalopathy within 48 hours
* Females - pregnancy, less than 12 weeks postpartum, lactating or willingness/intention to become pregnant during the study and for 3 months following vaccination.
* Seropositive for hepatitis B surface antigen (HBsAg) or Hepatitis C (antibodies to hepatitis C virus)
* Significant abnormal finding (in the setting of VL, see definitions in Inclusion criteria) on entry biochemistry or haematology blood tests or urinalysis
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* Tuberculosis, leprosy, or malnutrition (malnutrition in adults defined as a BMI <18.5, and in adolescents (12-17yrs) as a Z score cut-off value of <-2 SD).
* Any other significant disease, disorder or finding, which, in the opinion of a medically qualified Clinical Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Unlikely to comply with the study protocol

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety of single dose vaccination with ChAd63-KH | 12 months from vaccination
  Treatment-related adverse events as defined in the clinical trial protocol (median no. events)
Efficacy of single dose vaccination with ChAd63-KH | 12 months from vaccination
  Frequency of occurrence of PKDL in patients completing treatment with SSG / PM.

SECONDARY OUTCOMES:
Immunological response: T cells | 12 months from vaccination
  To compare systemic immune responses in vaccine vs placebo arms by measurement of the frequency (median) of gamma-interferon producing T cells
Immunological response: transcriptomics | 12 months from vaccination
  Comparing transcripts for differential expression in vaccine and placebo arms
Pathogenesis of PKDL comparing Leishmania parasite load pre-vaccination and at PKDL onset | 12 months from vaccination
  Parasite detection using RNAscope / immunocytochemistry
Immunological response: B cells | 12 months from vaccination
  Measurement of frequency in vaccinated and placebo groups of B cells by flow cytometry
Immunological response: antibody levels | 12 months from vaccination
  To compare systemic immune responses in vaccine vs placebo arms by median optical density levels

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Kaye, PhD, Study Director — University of York

IPD SHARING:
Plan to Share IPD: No